CLINICAL TRIAL: NCT02351557
Title: Effect of Cardiac Output on Uptake of Isoflurane
Brief Title: Pharmacokinetic Study of Effect of Cardiac Output on the Uptake of Isoflurane
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajarajan Ganesan, Junior Resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Other Study IDs: 9151/PG-2Trg/2012
Record Dates: First submitted 2015-01-16; First posted 2015-01-30 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Reference: Baseline cardiac index more than or equal to 2.1 liters per minute per square meter
- Low cardiac output: Baseline cardiac index less than 2.1 liters per minute per square meter

SUMMARY:
This study examines the effect of blood flow through the lungs and the body on the consumption and hence requirement of the anesthetic agent isoflurane.

DETAILED DESCRIPTION:
The effect of cardiac output on the uptake of isoflurane is yet to be quantified. This study aims to obtain a quantifiable relationship between isoflurane uptake and cardiac output. The study patients will be cardiac patients in whom anesthesia is induced with fentanyl , propofol and maintained on isoflurane . The baseline cardiac index from the pulmonary artery catheter as displayed on the continuous cardiac output monitor will be used to classify the patients into two groups with cardiac index of 2.1 liters per minute per square meter as the differentiating criteria. No change in the anesthesia protocol will be done for the two groups.The study is designed such that all vascular catheterisations and the dose of isoflurane administered is as per prevailing institutional protocols and that no other intervention particular or unique to the study is done. As such the data that the study will use is also routinely acquired during the procedure but not systematically stored, which is what the study will do. This, we suggest, makes the study an observational study.The continuous cardiac output data and the inspired and expired concentration of isoflurane as displayed on the monitor will be recorded online. Data will be collected from the start of isoflurane till 30 minutes or till the surgeon starts cannulating the great vessels. The data so obtained will be analysed in two groups based on the baseline cardiac index using Statistical Package for the Social Sciences (SPSS) for difference in uptake between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Presence of valve stenosis / valvular regurgitant lesion/ coronary artery disease with Ejection fraction >40%
* Posted for open cardiac surgery under general endotracheal anesthesia

Exclusion Criteria:

* Shunt lesion
* Allergy to propofol
* Psychotropic drug use
* Preinduction hemodynamic instability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing elective, open cardiac procedures under general endotracheal anesthesia with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Uptake of isoflurane in milliliter of vapor per minute | Every minute from 1 to 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: GOVERDHAN D PURI, MD,Ph.D, Study Director — Post Graduate Institute of Medical Education and Research, Chandigarh; Rajarajan Ganesan, M.D., Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Aveek Jayant, M.D.,D.M., Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Shyam Thingnam, M.S., Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

REFERENCES:
- [Background] Watt SJ, Cook LB, Ohri S, Lockwood GG. The relationship between anaesthetic uptake and cardiac output. Anaesthesia. 1996 Jan;51(1):24-8. doi: 10.1111/j.1365-2044.1996.tb07648.x. PMID 8669560
- [Background] Myles PS, Storer R, Millar C. Haemodynamic effects and uptake of enflurane in patients undergoing cardiac surgery: good versus poor myocardial function. Anaesth Intensive Care. 1992 Feb;20(1):21-7. doi: 10.1177/0310057X9202000104. PMID 1609936
- [Background] Kennedy RR, Baker AB. The effect of cardiac output changes on end-expired volatile anaesthetic concentrations--a theoretical study. Anaesthesia. 2001 Nov;56(11):1034-40. doi: 10.1046/j.1365-2044.2001.02212.x. PMID 11703234